CLINICAL TRIAL: NCT05923866
Title: A Phase 2, Double-blind, Placebo-controlled, Parallel-group Study Followed by an Open-label, Parallel Group Extension Part to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Potential Efficacy of Multiple Doses of ONO-2808 in Patients With Multiple System Atrophy
Brief Title: A Phase 2 Study of ONO-2808 in Patients With Multiple System Atrophy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONO-2808-03; jRCT2041230153 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-06-07; First posted 2023-06-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Multiple System Atrophy (MSA)
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ONO-2808 Arm (Experimental)
  Interventions: Drug: ONO-2808
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2808 — Oral administration of ONO-2808 at low, middle or high doses once a daily for 24 weeks
  Arms: ONO-2808 Arm
Drug: Placebo — Oral administration of placebo once a daily for 24 weeks
  Arms: Placebo Arm

SUMMARY:
This is a Phase 2, double-blind, parallel-group, placebo-controlled study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of multiple doses of ONO-2808 in patients with MSA. This is the first study of ONO-2808 in patients with MSA.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate 3 doses of ONO-2808 compared to placebo in MSA patients, including: 1) safety and tolerability, 2) pharmacokinetics, and 3) changes in clinical outcome assessments (COA) and biomarkers considered to be related to the pharmacodynamics and potential efficacy of ONO-2808.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients with a diagnosis of clinically-established or clinically-probable MSA according to the novel Movement Disorder Society (MDS) criteria for MSA diagnosis (2022), including patients with MSA of either subtype (MSA-P or MSA-C).
2. Patients at the early stages of the disease, defined as a maximum of 5 years since the onset of one of the following symptoms associated with MSA:

   * Parkinsonism
   * Ataxia
   * Orthostatic hypotension and/or urinary dysfunction
3. Patients with an anticipated survival of at least 3 years in the opinion of the Investigator.
4. Patients who are able to ambulate without the assistance of another person, defined as the ability to take at least 10 steps and then to turn around and walk at least another 10 steps. Use of assistive devices (e.g., walker or cane) is allowed.
5. Ability to swallow oral medication and be willing to adhere to the study intervention regimen.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Patients with a clinically-significant or unstable medical or surgical condition other than MSA that, in the opinion of the Investigator, might preclude safe completion of the study or might affect the results of the study (e.g., pulmonary, cardiovascular [including bradyarrhythmia], macular edema, and significant renal or hepatic dysfunction).
3. Neurological diseases/disorders other than MSA, such as Parkinson's disease, dementia with Lewy bodies, essential tremor, progressive supranuclear palsy, spinocerebellar ataxia, spastic paraparesis, corticobasal degeneration, or vascular, normal pressure hydrocephalus, pharmacological, or post-encephalitic parkinsonism.
4. Patients with documented liver diseases or cirrhosis.
5. Positive results at Screening for active viral infections that include positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) and hepatitis B core antibody, and hepatitis C virus (HCV).
6. Patients with suicide ideation according to the Investigator's clinical judgment per the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening or who have made a suicide attempt in the 6 months before Screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) | From screening up to follow-up (Week 28)
  Incidence of TEAEs, drug-related TEAEs, TEAEs resulting in study treatment discontinuation, TESAEs, and drug-related TESAEs will be tabulated by system organ class (SOC), preferred term (PT), and severity.
Vital signs (blood pressure) | From screening up to follow-up (Week 28)
  Summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
Vital signs (pulse rate) | From screening up to follow-up (Week 28)
  Summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
Vital signs (temperature) | From screening up to follow-up (Week 28)
  Summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
Vital signs (respiratory rate) | From screening up to follow-up (Week 28)
  Summaries of clinically significant and non-clinically significant abnormalities will be provided by each time point.
12-lead electrocardiograms (ECGs); parameters such as, but not limited to, heart rate, RR, PR, QRS, QT, and corrected QT intervals (QTcF) | From screening up to follow-up (Week 28)
  The number of patients with normal, abnormal not clinically significant and abnormal clinically significant of ECG results will be tabulated at each time point.
Clinically-significant abnormal physical examination findings | From screening up to follow-up (Week 28)
  The number of patients with normal, abnormal not clinically significant and abnormal clinically significant of physical examination results will be tabulated at each time point.
Clinical laboratory abnormalities (hematology, clinical chemistry, and urinalysis) | From screening up to follow-up (Week 28)
  The number of patients with abnormal laboratory results at any time during the study will be tabulated.
Clinically-abnormal findings in the Columbia Suicide Severity Rating Scale (C-SSRS) | From screening up to follow-up (Week 28)
  Responses to the suicidality assessment scale (C-SSRS) will be listed.

SECONDARY OUTCOMES:
Plasma concentration of ONO-2808 | Week 2, Week 8, Week 12, and Week 24
  Descriptive summary statistics will be calculated for ONO-2808 plasma concentrations, by dose level and time point.
ONO-2808 concentration in cerebrospinal fluid (CSF) | Week 24
  Descriptive summary statistics will be calculated for ONO-2808 CSF concentrations, by dose level and time point.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (35):
- United States (30):
  - The Parkinson's Movement and Disorder Institute, Fountain Valley, California
  - University of Southern California, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Yale School of Medicine - Yale Church Street Research Unit (CRSU), New Haven, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Norman Fixel Institute for Neurological Diseases - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan School of Medicine, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health - NYU Dysautonomia Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Penn State University - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The University of Pennsylvania - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Evergreen Health, Kirkland, Washington
  - Swedish Neuroscience Institute, Movement Disorders Clinic, Seattle, Washington
- Japan (5):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - National Hospital Organization Sendai Nishitaga Hospital, Sendai, Miyagi
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka, Osaka
  - Tokyo Metropolitan Neurological Hospital, Fuchū, Tokyo
  - National Hospital Organization Utano National Hospital, Kyoto

IPD SHARING:
Plan to Share IPD: No